CLINICAL TRIAL: NCT02740608
Title: An Open Label, Non-randomised, Prospective, Single Arm, 2-part Trial, Using Normothermic Machine Liver Perfusion NMLP to Test Viability and Transplantation of Marginal Livers
Brief Title: Viability Testing and Transplantation of Marginal Livers
Acronym: VITTAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Wellcome Trust (Other); University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG_15_240; 2016-001250-18 (EudraCT Number)
Record Dates: First submitted 2016-04-12; First posted 2016-04-15 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Liver transplantation (Other): All Participants will receive liver transplantation using the OrganOx metra device
  Interventions: Device: OrganOx metra

INTERVENTIONS:
Device: OrganOx metra — Normothermic Machine Liver Perfusion

SUMMARY:
This study is designed to determine if a rejected liver is viable using normothermic machine liver perfusion (NMLP). It aims to

1. establish the suitability of livers which have been declined by all UK liver transplant centres by monitoring their function on the NMLP machine; and,
2. transplant the liver if its function on the machine is satisfactory allowing it to be transplanted.

DETAILED DESCRIPTION:
Deaths from liver disease have soared by 40 per cent in a decade and continue to rise. Liver transplantation is a highly successful treatment of end stage liver disease, fulminant hepatic failure and early stage primary liver cancer. The demand for donor livers for transplantation greatly exceeds supply and approximately 20% of patients die whilst awaiting transplantation. Normothermic machine liver perfusion (NMLP) is a novel technique developed for the purposes of organ preservation, which we have also found allows monitoring of liver graft function ex-vivo by measuring bile production, whilst permitting objective assessment of liver biochemistry and blood flow. The OrganOx metra, the NMLP device we are using, is CE marked but is not currently licensed for this particular use and the livers will not be transported using this device (which the CE mark currently covers). The device will be used at a particular site (in this case University Hospitals Birmingham) and after a period of static cold storage during which the liver will be transported to the hospital for testing on the device. The study population will be extended criteria donor livers, rejected for transplantation by all UK centres, which are then found to be functioning during perfusion and transplanted into "medium to low-risk" liver transplant recipients. VITTAL is an open label, non-randomised, prospective, single arm, 2-part trial the objectives of which are to:

* Further validate liver viability assessment criteria
* Perform the phase 2 study transplanting successfully resuscitated "rejected" livers
* Establish the feasibility of NMLP as a means to increase the number of transplantable livers.
* Identify novel biomarkers that are indicative of liver quality and function In terms of intervention, the procurement and transplantation of the organs will follow the current standard of care. The only deviation from the current standard will be the normothermic perfusion of organs following static cold storage in order to test their ability to function. This study is based on results from a 5-case pilot series which transplanted low-risk recipients with organs that had been rejected for transplantation but had been shown to function on the normothermic machine perfusion device. This work is currently in the process of being published. The main risk would be the transplantation of a non-functioning graft (resulting in a case of primary non-function that could result in re-transplantation or patient death.) Based on our pre-clinical research and clinical pilot series we believe the criteria we have identified that indicate organ function are stringent and significantly reduce this risk.

ELIGIBILITY:
Inclusion Criteria (for the donor graft):

1. Liver from a donor primary accepted with the intention for a clinical transplantation
2. Liver graft was rejected by all the other UK transplant centres via normal or fast-track sequence
3. Cold ischaemic time less than 16 hours for DBD and 10 hours for DCD grafts
4. One of the following parameters capturing the objectivity of the liver high-risk status

   * Donor risk index greater than 2.0
   * Graft steatosis greater than 30%
   * BAR score greater than 9;
   * Donor warm ischaemic time greater than 30 minutes
   * Anticipated cold ischaemic time greater than 12 hours for DBD or 8 hours for DCD liver grafts
   * Suboptimal liver graft perfusion documented by a photo of macroscopic appearance
   * Liver transaminases (ALT or AST) above 1000 IU/mL

Exclusion Criteria (for the donor graft):

1. Grafts from patients with active Hepatitis B, C or HIV infection
2. Livers with cirrhotic macroscopic appearance
3. Livers with advanced fibrosis
4. DCD grafts with donor warm ischaemic time (systolic blood pressure less than 50mmHg to aortic perfusion) more than 60 minutes
5. Excessive cold ischaemic times (DBD more than 16 hours / DCD more than 10 hours)

Criteria for transplantation:

1. Evidence of bile production
2. Perfusate lactate levels less than or equal to 2.5 mmol/L 3. pH greater than 7.30

4. Metabolism of glucose 5. Stable arterial flow of more than 150 mL/ minute and portal flow more than 500 mL/minute 6. Homogeneous graft perfusion with soft consistency of the parenchyma

Inclusion Criteria (subject):

1. Adult primary liver transplant recipient
2. Patient listed electively for transplantation
3. Low to moderate transplant risk candidate, suitable for marginal graft, as assessed by the UHB liver transplant listing MDT meeting (these are usually candidates with low UKELD score, without cardiovascular comorbidities, with good functional and nutrition status, with patent portal vein and with no history of previous major upper abdominal surgery, e.g. patients transplanted for liver cancer)

Exclusion Criteria (subject):

Subjects who meet any of the following exclusion criteria are excluded from participating in the VITTAL trial:

1. High-risk patients and recipients not suitable for a marginal graft (these are mainly patients with high UKELD score (>62 as per the NHSBT LAG criteria for graft sharing in highrisks recipients in the North East of the UK [http://www.odt.nhs.uk/pdf/advisory.../Liver_National_Allocation_Scheme.pdf]), with cardiovascular comorbidities or renal insufficiency, with poor nutrition and performance status or history of major upper abdominal surgery, e.g. patients listed for liver re-transplantation)
2. Patients with complete portal vein thrombosis diagnosed prior to the transplantation
3. Liver re-transplantation
4. Patients with fulminant hepatic failure
5. Patients undergoing transplantation of more than one organ
6. Contraindication to magnetic resonance imaging (i.e. pacemaker fitted)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2018-05-08 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Patient survival | 90 days
  Achievement of successful transplantation of previously rejected donor liver following viability testing using NMLP
Use of NMLP to identify the proportion of transplantable liver grafts from the currently rejected donor organ pool. | Approximately 6 hours
  Decision point of using graft in patient transplantation

SECONDARY OUTCOMES:
Liver graft function | 12 month
  Assess the liver graft function following transplantation (by incidence of primary non-function, and early allograft dysfunction) by
  * Liver function tests
  * 90-day graft survival
  * 12-month patient and graft survival The secondary endpoints and other outcome measures will be compared with a contemporary matched recipient group
Morbidity associated with receipt of extended criteria graft | 90 days
  Assess morbidity associated with receipt of extended criteria graft that had previously been rejected by
  * Adverse event rates and severity
  * Requirement of renal replacement therapy
  * Incidence of biliary complications
  * Incidence of vascular complications
  * Biopsy-proven acute rejection
  * Reoperation rate
  * Length of intensive therapy unit stay
  * Length of hospital stay
Physiological response to reperfusion of the perfused grafts | Approximately 6 hours
  Assess the physiological response to reperfusion of the perfused grafts by
  • Post-reperfusion syndrome (Defined as a decrease in mean arterial pressure (MAP) of more than 30% from the baseline value for more than one minute during the first five minutes after reperfusion (assessed in the context of inotrope use)

CONTACTS AND LOCATIONS:
Overall Officials: Darius Mirza, Principal Investigator — University Hospital Birmingham NHS Foundation Trust
Locations (1):
- UHBFT - Queen Elizabeth Hospital, Birmingham, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laing RW, Mergental H, Yap C, Kirkham A, Whilku M, Barton D, Curbishley S, Boteon YL, Neil DA, Hubscher SG, Perera MTPR, Muiesan P, Isaac J, Roberts KJ, Cilliers H, Afford SC, Mirza DF. Viability testing and transplantation of marginal livers (VITTAL) using normothermic machine perfusion: study protocol for an open-label, non-randomised, prospective, single-arm trial. BMJ Open. 2017 Nov 28;7(11):e017733. doi: 10.1136/bmjopen-2017-017733. PMID 29183928
- [Background] Mergental H, Laing RW, Hodson J, Boteon YL, Attard JA, Walace LL, Neil DAH, Barton D, Schlegel A, Muiesan P, Abradelo M, Isaac JR, Roberts K, Perera MTPR, Afford SC, Mirza DF. Introduction of the Concept of Diagnostic Sensitivity and Specificity of Normothermic Perfusion Protocols to Assess High-Risk Donor Livers. Liver Transpl. 2022 May;28(5):794-806. doi: 10.1002/lt.26326. Epub 2021 Nov 9. PMID 34619014
- [Background] Mergental H, Laing RW, Afford SC, Mirza DF. Reply to 'Hypothermic machine perfusion before viability testing of previously discarded human livers'. Nat Commun. 2021 Feb 12;12(1):1015. doi: 10.1038/s41467-021-21183-7. No abstract available. PMID 33579911
- [Background] Neil DAH, Mergental H, Hann A, Laing RW, Hartog H, Mirza DF, Perera MTPR. Is Hepatocyte Necrosis a Good Marker of Donor Liver Viability During Machine Perfusion? Hepatol Commun. 2022 Feb;6(2):435-436. doi: 10.1002/hep4.1816. Epub 2021 Sep 2. No abstract available. PMID 34558864
- [Background] Attard JA, Osei-Bordom DC, Boteon Y, Wallace L, Ronca V, Reynolds G, Perera MTPR, Oo YH, Mergental H, Mirza DF, Afford SC. Ex situ Normothermic Split Liver Machine Perfusion: Protocol for Robust Comparative Controls in Liver Function Assessment Suitable for Evaluation of Novel Therapeutic Interventions in the Pre-clinical Setting. Front Surg. 2021 Feb 17;8:627332. doi: 10.3389/fsurg.2021.627332. eCollection 2021. PMID 33681282
- [Result] Mergental H, Laing RW, Kirkham AJ, Perera MTPR, Boteon YL, Attard J, Barton D, Curbishley S, Wilkhu M, Neil DAH, Hubscher SG, Muiesan P, Isaac JR, Roberts KJ, Abradelo M, Schlegel A, Ferguson J, Cilliers H, Bion J, Adams DH, Morris C, Friend PJ, Yap C, Afford SC, Mirza DF. Transplantation of discarded livers following viability testing with normothermic machine perfusion. Nat Commun. 2020 Jun 16;11(1):2939. doi: 10.1038/s41467-020-16251-3. PMID 32546694
- [Derived] Mergental H, Laing RW, Kirkham AJ, Clarke G, Boteon YL, Barton D, Neil DAH, Isaac JR, Roberts KJ, Abradelo M, Schlegel A, Dasari BVM, Ferguson JW, Cilliers H, Morris C, Friend PJ, Yap C, Afford SC, Perera MTPR, Mirza DF. Discarded livers tested by normothermic machine perfusion in the VITTAL trial: Secondary end points and 5-year outcomes. Liver Transpl. 2024 Jan 1;30(1):30-45. doi: 10.1097/LVT.0000000000000270. Epub 2023 Dec 15. PMID 38109282